CLINICAL TRIAL: NCT00633074
Title: Non-inferiority Study of GlaxoSmithKline Biologicals' Influenza Vaccine GSK576389A Using Different Formulations.
Brief Title: Non-inferiority Study of GSK Biologicals' Influenza Vaccine GSK576389A Using Different Formulations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111454
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Thiomersal-free FluAS25 adjuvanted vaccine group (Experimental): Subjects received 1 dose of thiomersal-free FluAS25 adjuvanted vaccine
  Interventions: Biological: Thiomersal-free FluAS25 adjuvanted vaccine (GSK576389A)
- Thiomersal reduced FluAS25 adjuvanted vaccine group (Experimental): Subjects received 1 dose of thiomersal reduced FluAS25 adjuvanted vaccine
  Interventions: Biological: Thiomersal reduced FluAS25 adjuvanted vaccine (GSK576389A)

INTERVENTIONS:
Biological: Thiomersal-free FluAS25 adjuvanted vaccine (GSK576389A) — Intramuscular administration, 1 dose
  Arms: Thiomersal-free FluAS25 adjuvanted vaccine group
Biological: Thiomersal reduced FluAS25 adjuvanted vaccine (GSK576389A) — Intramuscular administration, 1 dose
  Arms: Thiomersal reduced FluAS25 adjuvanted vaccine group

SUMMARY:
The purpose of this study is to show the non-inferiority of different formulations of GlaxoSmithKline Biologicials' influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female 65 years of age or older at the time of vaccination.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation (medical history and medical history directed examination) before entering into the study.

Exclusion Criteria:

* Suspected (based on clinical symptoms) or confirmed (based on laboratory results) influenza infection within the last 6 months.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 21 days after vaccination.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Previous vaccination against influenza with any seasonal vaccine since July 2007.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s) including egg and chicken protein.
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation (medical history and medical history directed physical examination) or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Any medical conditions in which IM injections are contraindicated

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 720 (Actual)
Dates: Start 2008-03-03; Primary Completion 2008-04-11 (Actual); Study Completion 2008-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Estonia (3):
  - GSK Investigational Site, Saku
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111454 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Started | 360 | 360
Completed | 359 | 360
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group | Total
Number analyzed (Participants) | 360 | 360 | 720
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72 (5.02) | 71.7 (4.88) | 71.85 (4.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 257 | 520
  Male | 97 | 103 | 200

OUTCOME MEASURES:

1. Primary Outcome: Serum Haemagglutination-inhibition (HI) Antibody Titer Against the Three Vaccine Strains
Description: Titers were expressed as Geometric Mean Titers (GMTs). The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: Days 0 and 21
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity including all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 357 | 360
Titer
  A/Solomon Islands [Day 0] | 6.0 [5.7 to 6.4] | 6.0 [5.7 to 6.3]
  A/Solomon Islands [Day 21] | 86.5 [75.8 to 98.8] | 93.1 [80.5 to 107.6]
  A/Wisconsin [Day 0] | 15.9 [13.9 to 18.1] | 14.9 [13.1 to 17.0]
  A/Wisconsin [Day 21] | 613.2 [540.1 to 696.1] | 519.3 [451.5 to 597.3]
  B/Malaysia [Day 0] | 13.2 [11.9 to 14.7] | 13.0 [11.7 to 14.5]
  B/Malaysia [Day 21] | 287.5 [255.9 to 323.1] | 264.9 [235.5 to 297.9]

2. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against the Three Vaccine Strains
Description: A seropositive subject was defined as a subject with a serum HI titer greater than or equal to 1:10. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 357 | 360
Subjects
  A/Solomon Islands [Day 0] | 67 | 62
  A/Solomon Islands [Day 21] | 342 | 338
  A/Wisconsin [Day 0] | 209 | 199
  A/Wisconsin [Day 21] | 357 | 359
  B/Malaysia [Day 0] | 215 | 208
  B/Malaysia [Day 21] | 355 | 357

3. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against the Three Vaccine Strains
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a four-fold increase in post-vaccination titer. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 357 | 360
Subjects
  A/Solomon Islands | 278 | 281
  A/Wisconsin | 336 | 337
  B/Malaysia | 332 | 335

4. Secondary Outcome: HI Antibody Seroconversion Factors
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 357 | 360
Fold increase
  A/Solomon Islands | 14.3 [12.6 to 16.3] | 15.6 [13.5 to 18.1]
  A/Wisconsin | 38.7 [33.6 to 44.5] | 34.8 [30.0 to 40.3]
  B/Malaysia | 21.8 [19.3 to 24.6] | 20.3 [18.0 to 22.9]

5. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against the Three Vaccine Strains
Description: A seroprotected subject was defined as a suject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 357 | 360
Subjects
  A/Solomon Islands [Day 0] | 10 | 6
  A/Solomon Islands [Day 21] | 280 | 287
  A/Wisconsin [Day 0] | 112 | 97
  A/Wisconsin [Day 21] | 350 | 348
  B/Malaysia [Day 0] | 74 | 75
  B/Malaysia [Day 21] | 349 | 351

6. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include ecchymosis, pain, redness and swelling. Any: any symptom regardless of intensity grade. Grade 3 pain: considerable pain at rest, which prevented normal everyday activities. Grade 3 ecchymosis, redness and swelling: more than 100 millimeter.
Time Frame: During a 7-day period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 360 | 360
Subjects
  Any ecchymosis | 7 | 6
  Grade 3 ecchymosis | 0 | 0
  Any pain | 237 | 246
  Grade 3 pain | 2 | 1
  Any redness | 152 | 161
  Grade 3 redness | 10 | 12
  Any swelling | 74 | 90
  Grade 3 swelling | 1 | 4

7. Secondary Outcome: Duration of Solicited Local Symptoms
Description: Duration was expressed as median number of days the symptom persisted. Solicited local symptoms assessed include ecchymosis, pain, redness and swelling.
Time Frame: During a 7-day period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort on those subjects who reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 237 | 246
Days
  Ecchymosis (N= 7; 6) | 4.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0]
  Pain (N= 237; 246) | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0]
  Redness (N= 152; 161) | 3.0 [1.0 to 7.0] | 4.0 [1.0 to 7.0]
  Swelling (N= 74; 90) | 3.5 [1.0 to 7.0] | 3.5 [1.0 to 7.0]

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, headache, myalgia, nausea, shivering and fever. Any: any symptom regardless of intensity grade; any fever: oral temperature greater than or equal to 38 degrees Celsius (°C). Grade 3: symptoms that prevented normal activity ; Grade 3 fever: oral temperature greater than 39°C. Related: symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 7-day period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 360 | 360
Subjects
  Any arthralgia | 78 | 87
  Grade 3 arthralgia | 1 | 2
  Related arthralgia | 75 | 85
  Any fatigue | 139 | 143
  Grade 3 fatigue | 2 | 0
  Related fatigue | 139 | 141
  Any headache | 109 | 107
  Grade 3 headache | 3 | 1
  Related headache | 109 | 105
  Any myalgia | 111 | 101
  Grade 3 myalgia | 1 | 3
  Related myalgia | 111 | 99
  Any nausea | 38 | 43
  Grade 3 nausea | 1 | 1
  Related nausea | 37 | 42
  Any shivering | 45 | 43
  Grade 3 shivering | 1 | 0
  Related shivering | 45 | 43
  Any fever | 34 | 38
  Grade 3 fever | 0 | 1
  Related fever | 34 | 38

9. Secondary Outcome: Duration of Solicited General Symptoms
Description: Duration was expressed as median number of days the symptom persisted. Solicited general symptoms assessed include arthralgia, fatigue, headache, myalgia, nausea, shivering and fever.
Time Frame: During a 7-day period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort on those subjects who reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 139 | 143
Days
  Arthralgia (N= 78; 87) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Fatigue (N= 139; 143) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Headache (N= 109; 107) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Myalgia (N= 111; 101) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Nausea (N= 38; 43) | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 6.0]
  Shivering (N= 45; 43) | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Fever (N= 26; 25) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 4.0]

10. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During a 21-day period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 360 | 360
Subjects
  Any AEs | 83 | 71
  Grade 3 AEs | 3 | 0
  Related AEs | 61 | 53

11. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: Medically Significant Conditions (MSCs) included all unsolicited adverse events that resulted in a medically attended visit.
Time Frame: During a 21-day period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 360 | 360
Subjects
  Any MSCs | 9 | 5
  Grade 3 MSCs | 3 | 0
  Related MSCs | 1 | 1

12. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (up to Day 21)
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Number analyzed (Participants) | 360 | 360
Subjects
  Any SAEs | 3 | 0
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Events collected by systematic assessment: 7-day follow-up period after vaccination. Events collected by non-systematic assessment: 21-day follow-up period after vaccination.
Arm/Group | Thiomersal-free FluAS25 Adjuvanted Vaccine Group | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group
Serious Adverse Events (participants affected / at risk) | 3/360 | 0/360
Other Adverse Events (participants affected / at risk) | 303/360 | 321/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thiomersal-free FluAS25 Adjuvanted Vaccine Group (N=360) | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group (N=360)
Arterial fibrillation (Cardiac disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thiomersal-free FluAS25 Adjuvanted Vaccine Group (N=360) | Thiomersal Reduced FluAS25 Adjuvanted Vaccine Group (N=360)
Pain (General disorders) | 237 | 246
Redness (General disorders) | 152 | 161
Swelling (General disorders) | 74 | 90
Arthralgia (General disorders) | 78 | 87
Fatigue (General disorders) | 139 | 143
Headache (General disorders) | 109 | 107
Myalgia (General disorders) | 111 | 101
Nausea (General disorders) | 38 | 43
Shivering (General disorders) | 45 | 43
Fever (General disorders) | 34 | 38
Injection site pruritus (General disorders) | 34 | 30
Injection site induration (General disorders) | 22 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.